CLINICAL TRIAL: NCT04286698
Title: To Investigate the Effectiveness of Two Different Physiotherapy Programs in Lymphedema Following Head and Neck Cancer Treatment
Brief Title: Two Different Physiotherapy Programs in Lymphedema Following Head and Neck Cancer Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Bakircay University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Kadirhan Ozdemir, PT, PhD., Head of Geriatric Rehabilitation Department, Izmir Bakircay University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2018-112
Record Dates: First submitted 2020-02-24; First posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Head and Neck Cancer; Lymphedema of Face; Fibrosis; Skin
Keywords: Complex decongestive physiotherapy; Home program; Manual lymph drainage; Face mask; 3D analysis
MeSH Terms: conditions — Head and Neck Neoplasms; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Complex decongestive physiotherapy program group (Active Comparator): Manuel lymph drainage, compression mask, exercises and skin care
  Interventions: Other: Complex decongestive physiotherapy
- Home program group (Active Comparator): Self-manuel lymph drainage and home exercises
  Interventions: Other: Home program
- Control group (No Intervention): No intervention

INTERVENTIONS:
Other: Complex decongestive physiotherapy — MLD was administered 5 days a week for 4 weeks, with each session lasting 30 minutes [25]. Compression therapy was applied to the patients by wearing a compression mask (FM Velcro Fastener, LIPOELASTIC), made of polyamide, cotton, viscose, and elastane, that covered the submandibular region, the masseter region, and the neck. The compression mask is specifically designed for the healing and recovery of tissues after plastic and aesthetic surgeries. The patients were advised to wear the compression masks for at least 4-6 hours per day for 4 weeks and gradually increase wearing time according to their tolerance. The patients were asked to perform skin care by themselves. Skin care was applied using a low pH skin lotion to moisturize the skin. Neck, face/mimic, tongue, and posture exercises were performed by patients while the compression mask was worn and under the supervision of a physiotherapist, with 10 repetitions 5 times a week for 4 weeks.
  Arms: Complex decongestive physiotherapy program group
Other: Home program — Self-MLD and exercises (neck, face/mimic, tongue, and posture exercises) were shown to the patients in this group. Self-MLD included self-administered lymph drainage of the axillary, posterior, lateral, and anterior neck areas; the pre- and retro-auricular regions; the lateral and anterior regions of the face; and the lower jaw region. Then the order is reversed back to the starting point [3]. A video of self-MLD and a text including exercise descriptions were shared with patients and their relatives to ensure that the self-MLD and exercises were performed accurately and regularly at home. Self-MLD was recommended to be applied once a day, and the exercises were advised to be performed for 10 repetitions each, 10 times a day for 4 weeks. The patients were called by phone during the second week after their first evaluation as a control and to motivate the patient for performing self-MLD and home exercises properly.
  Arms: Home program group

SUMMARY:
The aim of this study was to determine the effects of complex decongestive physiotherapy (CDP) and home programs on internal/external lymphedema, staging, fibrosis, and three-dimensional (3D) surface scanning and volume evaluation in head and neck lymphedema. Twenty-one patients were randomly divided into three groups: CDP; home program including self manual lymph drainage (MLD) and exercises; and control. CDP included MLD drainage, compression, exercise, and skin care. Self-MLD and exercises were performed by home program group patients. Assessment methods were applied at baseline and 4 weeks later for all groups. MD. Anderson Cancer Center Head and Neck Lymphedema Protocol was implemented to evaluate head and neck external lymphedema, staging, and fibrosis. An Artec Eva 3D scanner and the Autodesk ReCap Photo Studio software were used to determine and calculate the volume of the head and neck region via 3D surface scanning. Head and neck external lymphedema and fibrosis assessment criteria were performed to evaluate visible soft tissue edema and the degree of stiffness. To assess internal lymphedema, Patterson's scale was applied using fiber-optic endoscopic imaging.

DETAILED DESCRIPTION:
Head and neck cancer (HNC) have been seen in 13.3/100,000 males and 2.8/100,000 in females in Turkey. HNC related treatments such as lymph node dissection, tumor excision, chemotherapy, radiotherapy, and cancer itself can cause head and neck lymphedema (HNL). The incidence of HNL due to HNC treatments (surgery, chemotherapy and chemoradiation) has been reported to be between 48% and 90%.

A recognition of HNL has been growing in recent years, but HNL is still much less recognized than upper and lower limb lymphedema and is easily ignored by both patients and health care providers. Therefore, in many cases, the diagnosis and treatment of HNL may be delayed, or patients cannot access treatment. In routine practice, after HNC, the self-absorption of HNL is generally expected. Clinical experiences have confirmed that HNL develops 2-6 months after cancer treatment and regresses in some patients over time.

A variety of physiotherapy approaches have been shown to prevent and minimize physical, functional, emotional, and social disorders resulting from HNL. However, complex decongestive physiotherapy (CDP) is considered a gold standard treatment method for lymphedema. This method consists of manual lymph drainage (MLD), skin care, compression therapy, and therapeutic exercises. Although there are many studies about the effects of CDP on upper and lower limbs, there is only a limited number of studies about HNL and CDP in the literature.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* had unilateral/bilateral neck dissection
* had received radiotherapy and/or chemotherapy
* elapsed time of 3 or more months since cancer treatments
* had secondary HNL

Exclusion Criteria:

* having metastases due to HNC or other primary cancers
* receiving/having received treatment to regulate the lymph flow
* having the diagnosis of neurological, orthopedic, or rheumatologic diseases that may cause circulation and movement in the head and neck region.

Ages: 22 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Internal Lymphedema at 4 weeks | At baseline and 4 weeks later
  Patterson's scale is the most comprehensive scale for evaluating internal HNL. It is a fiber-optic endoscopic imaging method applied by an otolaryngologist to assess the gaps in the pharynx and larynx with regard to edema. Also, 11 different structures (base of tongue, posterior pharyngeal wall, epiglottis, pharyngoepiglottic folds, aryepiglottic folds, interarytenoid space, cricopharyngeal prominence, arytenoids, false vocal folds, true vocal folds, anterior commissure) and two spaces (vallecula and pyriform sinus) are rated as normal, mild, moderate, or severe during the inspection [26].
Change from Baseline External Lymphedema at 4 weeks | At baseline and 4 weeks later
  The MD Anderson Cancer Center HNL standard evaluation protocol includes two facial circumference measurements and nine point-to-point tape measurements between the reference points on the face [27].
  Seven key facial measurements were totaled to form a composite facial score. In addition, composite neck score was obtained by performing circumference measurements from three different regions of the neck [27].
  In order to clinically determine the development of external HNL, a reduction in the lymphedema stage or a minimum 2% reduction was required in absolute values in composite measurements that were equivalent to a change of at least 2 cm [2, 28].
Change from Baseline Staging Lymphedema at 4 weeks | At baseline and 4 weeks later
  The MD Anderson Cancer Center HNL rating scale was based on the traditional Földi's scale, which is used for staging limb lymphedema and determining the severity [3]. The only difference between the MD Anderson Cancer Center HNL rating scale and Földi's scale is that Stage 1 is divided into Stage 1a and Stage 1b on Földi's scale. Stage 0 demonstrates lymphedema without visible edema but with a complaint of tissue heaviness. Stage 1a represents soft visible edema without pitting and which is reversible. Stage 1b shows soft pitting edema, which remains reversible. Stage 2 displays firm pitting edema, which is irreversible but lacks tissue changes. Stage 3 lymphedema, the most severe of all stages, represents irreversible tissue changes such as hyperkeratosis or papillomatosis [27].
Change from Baseline Characteristics of Tissue Changes (edema and/or fibrosis), The Anatomical Locations, and The Severity of The Identified Soft Tissue Abnormalities at 4 weeks | At baseline and 4 weeks later
  The HNC related external lymphedema and fibrosis assessment criteria were used to evaluate the parameters, including the presence of visible soft tissue edema, the degree of stiffness of the tissues involved, and the severity of the lymphedema on the left periorbital region, right periorbital region, left cheek, right cheek, and submental region. This scale was used for rating the tissue under four headings for each region: Type A, Type B, Type C, and Type D. Next, each type other than Type A was graded as mild, moderate, and severe [29].
Change from Baseline 3D Surface Scanning and Volume Evaluation at 4 weeks | At baseline and 4 weeks later
  This evaluation was applied with an Artec Eva 3D scanner. The measurements and analyses were performed for seven different anatomical reference points. Seven markers were used to facilitate the calculation of the volume of the face and neck following the 3D scanning of the face and neck area; the data obtained were transferred to computer. After the scan was completed, a pattern atlas was created using the Autodesk ReCap photo software for the data on image, geometry, and texture. Finally, the predetermined reference points were combined, and the volume of the remaining portion was calculated by the volume of the 3D network representing the scanned geometry. In addition, the properties of the object were calculated using MESHLAB software.

CONTACTS AND LOCATIONS:
Locations (1):
- Kadirhan Ozdemir, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Smith BG, Hutcheson KA, Little LG, Skoracki RJ, Rosenthal DI, Lai SY, Lewin JS. Lymphedema outcomes in patients with head and neck cancer. Otolaryngol Head Neck Surg. 2015 Feb;152(2):284-291. doi: 10.1177/0194599814558402. Epub 2014 Nov 11. PMID 25389318
- [Background] Deng J, Ridner SH, Dietrich MS, Wells N, Wallston KA, Sinard RJ, Cmelak AJ, Murphy BA. Prevalence of secondary lymphedema in patients with head and neck cancer. J Pain Symptom Manage. 2012 Feb;43(2):244-52. doi: 10.1016/j.jpainsymman.2011.03.019. Epub 2011 Jul 30. PMID 21802897
- [Background] Ridner SH. Pathophysiology of lymphedema. Semin Oncol Nurs. 2013 Feb;29(1):4-11. doi: 10.1016/j.soncn.2012.11.002. PMID 23375061
- [Background] Deng J, Ridner SH, Murphy BA. Lymphedema in patients with head and neck cancer. Oncol Nurs Forum. 2011 Jan;38(1):E1-E10. doi: 10.1188/11.ONF.E1-E10. PMID 21186146
- [Background] Della Justina, L.B. and M. Dias, Head and neck lymphedema: what is the physical therapy approach? A literature review. Fisioterapia em Movimento, 2016. 29(2): p. 411-419.
- [Background] Smile TD, Tendulkar R, Schwarz G, Arthur D, Grobmyer S, Valente S, Vicini F, Shah C. A Review of Treatment for Breast Cancer-Related Lymphedema: Paradigms for Clinical Practice. Am J Clin Oncol. 2018 Feb;41(2):178-190. doi: 10.1097/COC.0000000000000355. PMID 28009597
- [Background] Watanabe Y, Koshiyama M, Seki K, Nakagawa M, Ikuta E, Oowaki M, Sakamoto SI. Development and Themes of Diagnostic and Treatment Procedures for Secondary Leg Lymphedema in Patients with Gynecologic Cancers. Healthcare (Basel). 2019 Aug 27;7(3):101. doi: 10.3390/healthcare7030101. PMID 31461980
- [Background] Crane P, Feinberg L, Morris J. A multimodal physical therapy approach to the management of a patient with temporomandibular dysfunction and head and neck lymphedema: a case report. J Man Manip Ther. 2015 Feb;23(1):37-42. doi: 10.1179/2042618612Y.0000000021. PMID 26309380
- [Background] Piso DU, Eckardt A, Liebermann A, Gutenbrunner C, Schafer P, Gehrke A. Early rehabilitation of head-neck edema after curative surgery for orofacial tumors. Am J Phys Med Rehabil. 2001 Apr;80(4):261-9. doi: 10.1097/00002060-200104000-00006. PMID 11277132
- [Background] Doke KN, Bowman L, Shnayder Y, Shen X, TenNapel M, Thomas SM, Neupane P, Yeh HW, Lominska CE. Quantitative clinical outcomes of therapy for head and neck lymphedema. Adv Radiat Oncol. 2018 Apr 27;3(3):366-371. doi: 10.1016/j.adro.2018.04.007. eCollection 2018 Jul-Sep. PMID 30202804
- [Derived] Ozdemir K, Keser I, Duzlu M, Erpolat OP, Saranli U, Tutar H. The Effects of Clinical and Home-based Physiotherapy Programs in Secondary Head and Neck Lymphedema. Laryngoscope. 2021 May;131(5):E1550-E1557. doi: 10.1002/lary.29205. Epub 2020 Oct 28. PMID 33111977